CLINICAL TRIAL: NCT05117541
Title: Bio-Psycho-Social Drivers of Disparities in Liver Disease Progression Among Korean Americans With Hepatitis B Infection
Brief Title: Social-environmental, Psychosocial, Behavioral, Clinical and Biological Drivers of Disparities in Liver Disease Progression Among Korean American With Chronic Hepatitis B Infection
Status: Active, not recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 21F.415; JT 17047 (Other: JeffTrial Number); R01DK125541 (NIH)
Record Dates: First submitted 2021-09-21; First posted 2021-11-11 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Chronic Viral Hepatitis; Hepatitis B Infection
MeSH Terms: conditions — Hepatitis B | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (interview, biospecimen collection): Patients participate in interviews over 20-40 minutes and undergo collection of hair samples at baseline and 18-24 months. Patients' medical records are also reviewed.
  Interventions: Other: Interview; Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Other: Interview — Participate in interviews
Procedure: Biospecimen Collection — Undergo collection of hair samples
Other: Electronic Health Record Review — Medical records are reviewed

SUMMARY:
This study explores how psychosocial factors (e.g., chronic stress, depression) may lead to liver disease progression such as liver cirrhosis or liver cancer among Korean American chronic hepatitis B infection patients. Gathering health information over time from Korean Americans with chronic hepatitis B infection may help doctors find better methods of treatment and on-going care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the prevalence of chronic hepatitis B (CHB) phenotype and liver disease severity at enrollment visit, and model how multiple social-environmental, psychosocial, behavioral, clinical and biological attributes are associated with variation in CHB phenotype and disease severity.

II. To identify how these same attributes are associated with disease progression over time.

SECONDARY OBJECTIVE:

I. To examine the moderating effects of these multi-level factors on the relationship between liver disease progression and adverse liver disease outcome (e.g., hepatocellular carcinoma [HCC]), as well as mediating effects of liver disease progression on the relationship between psychosocial factors and liver cancer or death.

EXPLORATORY OBJECTIVE:

I. Using an explanatory mixed methods approach, to understand the care-seeking behaviors, and dynamics of care, within an ethnically concordant liver disease care model, and how these factors may have both direct and mediational effects on adherence, treatment effectiveness, and adverse disease outcomes.

OUTLINE:

Patients participate in interviews over 20-40 minutes and undergo collection of hair samples at baseline and 18-24 months. Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Korean-American male or female, age over 18 and older
* CHB Patients who have lab and medical record data (including hepatitis B virus [HBV] deoxyribonucleic acid [DNA] viral load, hepatitis B virus e Antigen [HBeAg] status, and liver enzyme values) exist from 2015 or before

Exclusion Criteria:

* Patients who have received a diagnosis of HCC, although they may have been diagnosed with cirrhosis
* Patients who have been diagnosed with other viral infections (hepatitis C virus [HCV], human immunodeficiency virus [HIV], etc.)
* Patients who have total baldness

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Korean American patients with chronic hepatitis B infection at Liver Disease Prevention Center, Thomas Jefferson University Hospital (TJUH) or Asian Pacific Liver Center (APLC), Coalition of Inclusive Medicine
Sampling Method: Non-Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change Chronic hepatitis B (CHB) phenotype | At start of treatment
  Categorized as follows: 1) immune tolerant, 2) immune active with hepatitis B virus e antigen (HBeAg)(+), 3) immune active with HBeAg(-), and 4) inactive carrier, with patients not fitting into one of these four phenotypes classified as 5) indeterminant. Phenotype at study enrollment will be calculated
Change Liver disease severity | At end of treatment
  Will be estimated using fibrosis 4 (FIB-4) (a parameter calculated using alanine aminotransferase [ALT] and aspartate aminotransferase [AST] values, platelet count and age) and APRI (AST to platelet ratios).

SECONDARY OUTCOMES:
Change in hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels | Baseline to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States